CLINICAL TRIAL: NCT02798341
Title: The Breast Program - Translational Cancer Resource
Acronym: TRACR
Status: Active, not recruiting | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: UPCC 08110
Record Dates: First submitted 2016-06-09; First posted 2016-06-14 (Estimated); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor Tissue Healthy Tissue Buffy Coat DNA Plasma Serum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Biospecimen Collection

SUMMARY:
TRACR will provide a data/biospecimen repository for translational research to better diagnose, prognose, treat and cure breast cancer (and related diseases/treatment conditions). Patients at the Rowan Breast Center will be consented for donation of blood and if available tumor/healthy/archived tissue. Patients will be consented to give permission to use said specimens for future research and to be contacted in the future about other research participation and additional information.

ELIGIBILITY:
Inclusion Criteria:

* RBC patients with known invasive cancer pre-surgery (greater or equal to 1.5cm) are given priority in recruitment.
* RBC patients with known invasive cancer pre-surgery (less then 1.5cm). 3. RBC patients who are postsurgery for invasive breast cancer (performed at UPHS or non-UPHS entities).
* Patients that are of high risk for breast cancer (family history, known deleterious genetic mutation(s)) seeking a prophylactic mastectomy at the breast clinic.
* Only persons who can understand and give informed consent will be eligible to participate in this study. Furthermore, no persons belonging to vulnerable populations with as children (below 18 years of age), fetuses, neonates or prisoners will be recruited in this study. Pregnant women, who are pre-surgery and having surgery for clinical reasons, can still be recruited for tissue and blood collection.

Exclusion Criteria:

* Individual who cannot understand and give informed consent (cognitively impaired persons)
* Children (below 18 years of age), fetuses and neonates
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast Cancer
Sampling Method: Probability Sample
Enrollment: 4000 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Number of biospecimen collected | 15 years

CONTACTS AND LOCATIONS:
Overall Officials: Angela DeMichele, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States